CLINICAL TRIAL: NCT01719276
Title: EFFECT OF COGNITIVE-BEHAVIORAL THERAPY AND EXERCISE VERSUS SUPERVISED EXERCISE PROGRAM IN PATIENTS WITH CHRONIC PAIN LUMBAR NO SPECIFIC: RANDOMIZED CONTROLLED TRIAL
Brief Title: Graded Activity Versus Supervised Exercises in Patients With Chronic Non-specific Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Mauricio Oliveira Magalhães, Mauricio Oliveira Magalhães, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: mauriciomag20
Record Dates: First submitted 2012-10-26; First posted 2012-11-01 (Estimated); Last update posted 2014-06-16 (Estimated); Status verified 2014-06

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Graded Activity (Active Comparator): Exercise treadmill, Strengthening of the lower limbs and trunk
  Interventions: Other: Graded Activity; Other: Supervised Exercises
- Supervised exercises (Active Comparator): Stretching, Strengthening, Motor Control
  Interventions: Other: Graded Activity; Other: Supervised Exercises

INTERVENTIONS:
Other: Graded Activity — The graded activity program to increase activity tolerance by performing individualized and submaximal exercises.
Other: Supervised Exercises — The group will perform stretching exercises (gluteus maximus, hamstrings, triceps surae, lumbar paraspinal), strengthening muscles (rectus abdominus, obliques and lower rectus abdominis internal and external) and motor control exercises (muscle transversus abdominis and lumbar multifidus.

SUMMARY:
The purpose of this study is to compare the efficacy of graded activity program and supervised exercise on pain, functional disability, quality of life, global perceived effect, return to work, physical activity, physical capacity and strength of the lower limbs in patients with chronic non-specific low back pain

DETAILED DESCRIPTION:
Objective: To contrast the efficacy of of graded activity program and supervised exercise on pain, functional disability, quality of life, global perceived effect, return to work, physical activity, physical capacity and strength of the lower limbs in patients with chronic non-specific low back pain

Design: Sixty-six will be randomized into two groups namely: Graded Activity program (GA)(n = 33) and supervised exercise (SE) (n = 33). The primary clinical outcomes will be pain, assessed with the numerical pain scale and McGill Pain Questionnaire, and disability assessed with Roland Morris Disability Questionnaire. Secondary outcomes will be measured with Global Perceived Effect, quality of life, return to work, physical activity, functional capacity and strength of the lower limbs. The program lasts for 6 weeks, and sessions happen twice a week, with duration of one hour each. Evaluations will be performed before(baseline), after (6weeks) and with a follow-up 3 and 6 months after treatment. Data will be collected by a blinded examiner who also had made the allocation of patients to groups. Significance level is established at 5%.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-specific chronic low back pain for at least three months, age between 18 and 65 year of both genders and with a minimum pain intensity score of three in the 11-point Pain Numerical Rating Scale (ranging from 0 to 10 points).

Exclusion Criteria:

* Known or suspected serious spinal pathology (fractures, tumors, inflammatory or infective diseases of the spine);

  * Nerve root compromise;
  * Comorbid health conditions that would prevent active participation in the exercise programs;
  * Pregnancy;
  * Cardio Respiratory illnesses;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2013-02; Primary Completion 2014-01 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Pain | 6 weeks
  Pain Numerical Rating Scale (NRS) and McGill Pain Questionnaire
Functional Disability | 6 weeks
  Roland Morris Disability Questionnaire

SECONDARY OUTCOMES:
Quality of life | 6 weeks
  Short-Form Health Survey Questionnaire
Global Perceived Effect | 6 weeks
  Global Perceived Effect Scale
Return to work | 6 weeks
  Patients will be asked if returned their professional activities.
Habitual physical activity | 6 weeks
  The Baecke questionnaire on habitual physical activity
Physical Capacity | 6 weeks
  physical capacity tests (sit-to-stand and 50-foot walk)
Kinesiophobia | Tampa Scale of Kinesophobia (TSK)
  self-applied questionnaire consisting of 17 items, which was developed to measure the fear of movement due to cLBP. Each question has 4 response options (strongly disagree, disagree, agree, and strongly agree) with scores respectively ranging from 1 to 4 points.

CONTACTS AND LOCATIONS:
Overall Officials: Amelia P Marques, PHD, Study Director — University of Sao Paulo; Mauricio O Magalhaes, MSc, Principal Investigator — University of Sao Paulo
Locations (1):
- Medicine School of the University Of São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Magalhaes MO, Franca FJ, Burke TN, Ramos LA, de Moura Campos Carvalho e Silva AP, Almeida GP, Yuan SL, Marques AP. Efficacy of graded activity versus supervised exercises in patients with chronic non-specific low back pain: protocol of a randomised controlled trial. BMC Musculoskelet Disord. 2013 Jan 21;14:36. doi: 10.1186/1471-2474-14-36. PMID 23336703